CLINICAL TRIAL: NCT02769559
Title: Reduction Mammaplasty Safely Increases the Quality of Life in Patients With Mammary Hypetrophy.
Brief Title: Reduction Mammaplasty and Improved Quality of Life
Acronym: MammaRed
Status: Completed | Type: Observational
Sponsor: University Hospital Bratislava (Other)
Collaborators: Comenius University (Other)
Responsible Party: Principal Investigator, Julius Hodosy, Reduction mammaplasty safely increases the quality of life in patients with mammary hypetrophy., University Hospital Bratislava
Other Study IDs: UHB/005/2015/MB
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Macromastia; Signs and Symptoms; Quality of Life
MeSH Terms: conditions — Gigantomastia; Signs and Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with macromasty: Female adult patients with symptomatic macromasty selected for elective reduction surgery
  Interventions: Procedure: Reduction mammaplasty

INTERVENTIONS:
Procedure: Reduction mammaplasty — Surgical removal of excess breast tissue

SUMMARY:
The data gathered here will be used to evaluate the efficacy and safety of the mammary reduction in patients with macromastia.

DETAILED DESCRIPTION:
The data was gathered using retrospective and follow-up prospective study of a group of patients, consisting of adult women that underwent a breast reduction surgery at the Clinic of Plastic, Reconstructive and Aesthetic Surgery Faculty of Comenius University and at the University Hospital in Bratislava, Ružinov, during the time period between 2000 until May 2014. The data concerning the quality of life of these patients was gathered by using the globally standardized questionnaire "Breast Q questionnaire©" with the separate software system evaluation tool "QScore©". The statistical analysis was conducted using GraphpadPrism program v. 6.01. The total number of respondents consisted of 52 people who were followed-up for up to 12 years.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years
* macromastia on clinical examination
* fulfilled Breast Q Questionnaire prior to surgery and after surgery
* signed informed consent

Exclusion Criteria:

* failed to sign informed consent
* failed to fill the Breast Q Questionnaire
* patients with altered mental status and behaviour
* patients with concomitant breast disease, or with previous breast interventions as are radiotherapy, surgery, or breast cancer

Ages: 18 Years to 63 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females with macromastia undergoing elective reduction surgery.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2000-01; Primary Completion 2014-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Quality of life | 2000-2014
  Questionnaires about quality of life before and up to 12 years after surgery

SECONDARY OUTCOMES:
Rate of adverse outcomes | 2000-2014
  Evaluation of rate and types of negative outcomes up to 12 years after elective reduction surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bratislava, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No